CLINICAL TRIAL: NCT00280956
Title: A Phase III, Multicenter, Open-Label, Long-Term Study of the Safety, Tolerability, and Efficacy of Intravenous Antegren™ (Natalizumab) in Crohn's Disease Subjects Who Have Previously Participated in Antegren Crohn's Disease Studies
Brief Title: Open Label Natalizumab Safety Extension Study for Subjects With Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CD351
Record Dates: First submitted 2006-01-21; First posted 2006-01-24 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Natalizumab

INTERVENTIONS:
Drug: natalizumab

SUMMARY:
The primary objective of this study is to evaluate the long-term tolerability and safety of natalizumab when administered a dose of 300 mg intravenously (IV) to subjects with Crohn's Disease who have previously participated in studies CD251, CD301, CD303, CD306, or CD307.

ELIGIBILITY:
* Male and Female Subjects 18 years and older with Crohn's Disease who have participated in studies CD251, CD301, CD303, CD306, or CD307 per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2002-07; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of natalizumab by the number and proportion of subjects with adverse events, and by assessing clinical laboratory parameters and vital signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Performed only at CD251, CD301, CD303, CD306, and CD307 sites globally. No general public enrollment. The study is managed from the office of Elan Pharmaceuticals, Inc. in, San Diego, California, United States